CLINICAL TRIAL: NCT05373810
Title: Registration Study on Bone and Soft Tissue Sarcoma - An Observational Cohort Study -
Brief Title: Registration Study Sarcoma
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Radiotherapiegroep (Other)
Responsible Party: Sponsor
Other Study IDs: NL69559.091.19
Record Dates: First submitted 2021-01-22; First posted 2022-05-13 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Surgical Procedures, Operative; Radiation; Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Surgery — all interventions are allowed
  Other Names: Radiation; Systemic treatment

SUMMARY:
The prospective and retrospective data collection on bone and soft tissue sarcoma is an observational cohort study aimed to collect clinical data and patient reported outcomes of all patients who have been diagnosed with bone or soft tissue sarcoma in the Netherlands. All patients diagnosed with bone or soft tissue sarcoma who are treated, planned for treatment or currently being treated, will be asked to participate in this project.

DETAILED DESCRIPTION:
The main objectives of this project are:

* To improve the knowledge and therefore the treatment care, in patients with bone or soft tissue sarcoma in the Netherlands
* To start an observational cohort study of bone and soft tissue sarcoma patients from their primary diagnosis until death
* To prospectively and retrospectively collect data on medical history, co-morbidities, baseline clinical parameters, imaging results, pathology results, tumor characteristics, treatment, treatment outcomes, functional outcome, cosmetic outcome, hospital stays and interventions.
* To collect data on health related quality of life and work ability, to collect data on patient reported outcomes measures.
* To create a continuous basis for a large variety of research purposes including:

  * Prognostic and predictive research
  * Health care policies and cost-effectiveness studies

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven bone or soft tissue sarcoma, excluding Gastrointestinal Stromal Tumours

Exclusion Criteria:

* Altered mental status that would prohibit the understanding of and giving of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with bone or soft tissue sarcoma who are recently diagnosed, currently under treatment or have been treated will be asked to participate in this cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2029-04-02 (Estimated); Study Completion 2029-04-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | up to 10 years
  PFS

SECONDARY OUTCOMES:
Health related quality of life | up to 5 years
  measured by EORTC QOL questionnaires
grade 3/4 serious adverse events | up to 5 years
  AE
Disease free survival | up to 10 years
  DFS
Overall survival | up to 10 years
  OS

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Radiotherapiegroep, Arnhem
  - Radboudumc, Nijmegen

IPD SHARING:
Plan to Share IPD: No